CLINICAL TRIAL: NCT00156338
Title: Effect of Intraoperative Fluid Management on Morbidity in Patients Undergoing Colorectal Surgery
Brief Title: Effect of Intraoperative Fluid Management on Morbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 02-Anast-05
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Epidural Anesthesia
Keywords: Fluid therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): volume and sodium restriction
  Interventions: Procedure: fluid management
- 2 (Active Comparator): volume restriction
  Interventions: Procedure: fluid management
- 3 (Active Comparator): liberal fluid management
  Interventions: Procedure: fluid management

INTERVENTIONS:
Procedure: fluid management — volume and sodium restriction
  Arms: 1
Procedure: fluid management — volume restriction
  Arms: 2
Procedure: fluid management — liberal fluid management
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether intraoperative fluid and sodium restriction decreases postoperative morbidity

ELIGIBILITY:
Inclusion Criteria:

* epidural anesthesia
* ASA I-III

Exclusion Criteria:

* metastasized cancer
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2005-07; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
all cause Morbidity | one year

SECONDARY OUTCOMES:
Gastral and intestinal function | within the first 30 days after surgery
all cause Mortality | one year
Gastral and intestinal function | one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Martin Westphal, MD, Principal Investigator — Department of Anesthesiology and Intensive Care, University Hospital Münster
Locations (3):
- Germany (3):
  - Raphaelsklinik, Münster
  - St. Franziskus-Hospital Münster, Münster
  - Department of Anesthesiology and Intensive Care, University Hospital Münster, Münster